CLINICAL TRIAL: NCT03640091
Title: Implant in Mandibular Molars
Brief Title: Pre-extractive Inter-radicular Implant Bed Preparation Versus Conventional Post-extractive Inter-radicular Implant Bed Preparation in Mandibular Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed abdel wahid elshoaby, Short implant, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cairo university 1
Record Dates: First submitted 2018-07-11; First posted 2018-08-21 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Randomized Clinical Trial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre-extractive inter-radicular implant bed preparation (Experimental)
  Interventions: Procedure: Post-extractive inter-radicular implant bed preparation

INTERVENTIONS:
Procedure: Post-extractive inter-radicular implant bed preparation — Implant placement in mandibular molars

SUMMARY:
Pre-extractive Inter-radicular Implant Bed Preparation versus Conventional Post-extractive Inter-radicular Implant Bed Preparation in Mandibular Molars

ELIGIBILITY:
Inclusion Criteria:

* Patients with badly decayed posterior molar teeth.
* Distance from height of inter-radicular furcation of mandibular molars to the mandibular canal should be equal to or more than 10 mm

Exclusion Criteria:

* Distance from height of inter-radicular furcation of mandibular molars to the mandibular canal equal to or less than 8 mm.
* Heavy smokers more than 20 cigarettes per day.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Implant stability | 1 year
  By ostell in newten scale

SECONDARY OUTCOMES:
Marginal bone loss | 1 year
  By cone beam xray in millimeters scale

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt